CLINICAL TRIAL: NCT03879889
Title: Smoking Reduction Intervention for Smoking Parents of Paediatric Patients in Hong Kong: a Randomised Controlled Trial
Brief Title: Smoking Reduction Intervention for Smoking Parents of Paediatric Patients in Hong Kong
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Kate Ching Ching Chan, Clinical Professional Consultant, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 01150077
Record Dates: First submitted 2019-03-13; First posted 2019-03-19 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Smoking, Tobacco
Keywords: Smoking reduction; Randomised controlled trial; Motivational interview; Nicotine replacement therapy; Environmental tobacco smoke exposure; Paediatrics; Children
MeSH Terms: conditions — Tobacco Smoking; Smoking Reduction | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Intervention Model Description: A single blinded randomized controlled trial aiming to evaluate the effectiveness of smoking reduction interventions for smoking parents in paediatric hospital setting in Hong Kong. This trial consists of a 24-week intervention period. Eligible families will be randomly assigned to either intervention group or control group. Smoking parent(s) in intervention group will be given face-to-face counselling on smoking reduction and adherence to nicotine replacement therapy (NRT) with motivational interviews, provision of NRT and monthly phone follow-up for counselling and support. Smoking parent(s) in control group will be given standard advice and information on smoking cessation.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Research study personnel who will conduct the data collection on outcome measures will be blinded to the group assignment. The researchers who will conduct the data analysis will also be blinded the group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Intervention arm will include face-to-face counseling on smoking reduction and adherence to nicotine replacement therapy (NRT) with motivational interviews, provision of free NRT, referral to quit smoking hotline, monthly phone follow-up and two follow-up visits.
  Interventions: Drug: Nicotine patch
- Control (No Intervention): Smoking parents will be given standard advice on smoking cessation. They will be given an information leaflet showing standard information on the currently available smoking cessation service as well as a smoking cessation hotline.

INTERVENTIONS:
Drug: Nicotine patch — Four weeks of nicotine patch will be provided at the first contact, which will be prescribed using the guidelines based on the subject's daily cigarette consumption. At week-4 visit, four more weeks of NRT will be provided.
  Other Names: Nicotinelle
  Arms: Intervention

SUMMARY:
A randomized controlled trial to evaluate the effectiveness of smoking reduction interventions for smoking parents in paediatric hospital setting in Hong Kong.

DETAILED DESCRIPTION:
This is a single blinded randomized controlled trial aiming to evaluate the effectiveness of smoking reduction interventions for smoking parents in paediatric hospital setting in Hong Kong. This trial consists of a 24-week intervention period. Eligible families will be randomly assigned to either intervention group or control group. Smoking parent(s) in intervention group will be given face-to-face counselling on smoking reduction and adherence to nicotine replacement therapy (NRT) with motivational interviews, provision of NRT and monthly phone follow-up for counselling and support. Smoking parent(s) in control group will be given standard advice and information on smoking cessation.

ELIGIBILITY:
Inclusion Criteria:

* Ethnic Chinese family with children aged younger than 18 years of age.
* Children who are admitted to the paediatric inpatient units or attend the paediatric specialist clinic at the Prince of Wales Hospital.
* Children with at least one custodial smoking parent who is living with them.
* Written informed consent obtained from parents.

Exclusion Criteria:

* Families not residing in Hong Kong.
* Children in foster care.
* Children with unclear custody.
* Smoking paediatric patients.
* Presence of smoking household members apart from the parents.
* Smoking parent who is contraindicated to use nicotine replacement therapy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Validated successful smoking reduction rate | Week-24
  Urinary cotinine validated parental successful smoking reduction rate at week-24
Self-reported parental successful smoking reduction rate at week-24 | Week-24
  Self-reported reduction of daily cigarette consumption by 50% or more compared with baseline

SECONDARY OUTCOMES:
Urinary cotinine validated parental smoking cessation rate at week-24 | Week-24
  Urinary cotinine validated parental smoking cessation rate at week-24
Parental self-reported smoking reduction rate of cigarette consumption | Week-24
  Parental self-reported smoking reduction rate of cigarette consumption
Parental self-reported smoking cessation rate of cigarette consumption | Week-24
  Parental self-reported 7-day point-prevalence tobacco abstinence
Change in children's urinary cotinine level from baseline to week-24 | Week-24
  Change in children's urinary cotinine level from baseline to week-24

CONTACTS AND LOCATIONS:
Overall Officials: Ching Ching Chan, FHKAM, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dai S, Chan MHM, Kam RKT, Li AM, Au CT, Chan KC. Monthly Motivational Interview Counseling and Nicotine Replacement Therapy for Smoking Parents of Pediatric Patients: A Randomized Controlled Trial. Front Pediatr. 2022 Apr 13;10:798351. doi: 10.3389/fped.2022.798351. eCollection 2022. PMID 35498786